CLINICAL TRIAL: NCT06883929
Title: The Effect of Vırtual Realıty Applıcatıon on the Anxıety and Fear Levels of Chıldren Who Are Planned for Daıly Surgery
Brief Title: The Effect of Virtual Reality Application on Anxiety and Fear Levels of Children Planned for Daily Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cihat Ozyılmaz (Other)
Responsible Party: Sponsor-Investigator, Cihat Ozyılmaz, Student, Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BİTLİS-HEM-CÖ-01
Record Dates: First submitted 2025-01-22; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Child; Fear; Anxiety
Keywords: Child; Anxiety; Fear; Distraction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Data Collection (Experimental): Equal numbers (n) (40:40) were included in the intervention and control groups by block randomization. Written informed consent was obtained from the parents and verbal consent was obtained from the children. Blood pressure and heart pulse was measured with the same calibrated devices throughout the study. The first and last measurements were evaluated by the researcher. In the intervention group five experts were consulted in order to involve children in the decision-making process. Three minutes and two six-minute video options. The videos show the forest, trees, flowers and 3D animated videos with animals and instrumental music were shown. Video maximum 30 minutes after being monitored. Both intervention and control group underwent the procedures to be applied in the preoperative period. The control group was not shown a video and only ward routines were applied.
  Interventions: Device: virtual reality glasses; Device: virtual reality goggles
- control group (No Intervention): Routine maintenance was provided

INTERVENTIONS:
Device: virtual reality glasses — Animation video application with virtual glasses by the researcher himself was applied. The application was performed in a quiet environment in the patient's room, in a sitting area where the child was comfortable.
  position and wearing virtual goggles over his eyes.
  Arms: Data Collection
Device: virtual reality goggles — vr 360 degree screen viewing
  Arms: Data Collection

SUMMARY:
Objective: This study was conducted to determine the effect of the animation video to be watched by child patients aged 5-10 before day surgery on their anxiety and fear levels in the preoperative period. Method: This research, which was conducted as a randomized controlled experimental study, was conducted with 80 children. Participants sociodemographic data, blood pressure, heart rate, Child Fear Scale and Yale Modified Preoperative Anxiety Scale Child Form were used to collect data. Comparisons in independent pair groups with Kolmogorov Smirnow Test whether the data received comply with normal distribution; Since the assumption of normality is met, comparisons in dependent pair groups are made with the significance test (t test) of the difference between two means; Since the assumption of normality was met, the significance test of the difference between two spouses was performed (two paired samples t test).

DETAILED DESCRIPTION:
Objective: This study was conducted to determine the effect of the animation video to be watched by child patients aged 5-10 before day surgery on their anxiety and fear levels in the preoperative period. Method: This research, which was conducted as a randomized controlled experimental study, was conducted with 80 children. Participants sociodemographic data, blood pressure, heart rate, Child Fear Scale and Yale Modified Preoperative Anxiety Scale Child Form were used to collect data. Comparisons in independent pair groups with Kolmogorov Smirnow Test whether the data received comply with normal distribution; Since the assumption of normality is met, comparisons in dependent pair groups are made with the significance test (t test) of the difference between two means; Since the assumption of normality was met, the significance test of the difference between two spouses was performed (two paired samples t test).

ELIGIBILITY:
Inclusion Criteria:

Not having an audiovisual disease

Exclusion Criteria:

Having an audiovisual disease

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Child fear scale | 6 months
  Child Fear Scale ranges from neutral (0 points=no fear) to frightened It consists of five different statements ranging up to one hundred (4 points=severe fear). Horror score the higher the level of fear, the higher the level of fear

SECONDARY OUTCOMES:
Yale modified preoperative anxiety scale pediatric form | 6 months
  In the scale consisting of four parts, points are evaluated all sections are scored within each section and the highest score in its section is divided by the grade. The scores from all sections are added up, divided by 4 again, and then divided by 100.
  is multiplied. This calculation results in a score between 22.92-100. High score refers to high anxiety and worry.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Il Sağlık Müdürlüğü, Bitlis, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No